CLINICAL TRIAL: NCT03792035
Title: China Tongxinluo Study for Myocardial Protection in Patients With Acute Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, fuwaihospital, Assistant dean, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-YFC-03-CTS-AMI; 2017YFC1700503 (Other Grant/Funding Number: National Key R&D Program-Research ; Modernization of TCM)
Record Dates: First submitted 2018-12-03; First posted 2019-01-03 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — tongxinluo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): First time given 8 capsules of Tongxinluo, then given 4 capsules of Tongxinluo, tid, po.Dosage form: capsule;Dose: 0.26g/capsule;Duration:1 year
  Interventions: Drug: Tongxinluo
- Control group (Placebo Comparator): First time given 8 capsules of placebo, then given 4 capsules of placebo, tid, po.Dosage form: capsule;Dose: 0.26g/capsule;Duration:1 year
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tongxinluo — tid, po.
  Arms: Experimental group
Drug: Placebos — tid, po.
  Arms: Control group

SUMMARY:
To determine the therapeutic effects of Tongxinluo Capsules as compared with placebo in the treatment of patients with acute ST-elevation myocardial infarction (STEMI): (1) Clinical efficacy and safety at 30 days: the incidence of composite endpoints comprising major adverse cardiovascular and cerebrovascular events (MACCE, including cardiovascular death, myocardial re-infarction, emergency coronary revascularization and cerebral stroke), severe complications (including cardiogenic shock, heart failure, mechanical complications and malignant arrhythmias), and major bleeding (BARC grade III and V); (2) Clinical efficacy and safety at 1 year: the incidence of composite endpoints comprising MACCE, hospitalization due to heart failure, in-stent thrombosis, and major bleeding (BARC grade III and V), as well as all-cause mortality; (3) the effects in promoting myocardial reperfusion, reducing incidence of myocardial no-reflow, protecting ischemic myocardium, minimizing infarction size, and improving left ventricular systolic function.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years;
2. Within 24 hours of infarctional chest pain onset;
3. ECG shows ST-segment elevation ≥0.2mV in more than 2 adjacent leads, or new left bundle branch block (LBBB);
4. Voluntary participation in the study with consent forms signed.

Exclusion Criteria:

1. Critically illness due to STEMI;
2. Long-term (>20 min) cardio-pulmonary resuscitation (CPR);
3. Suspected aortic dissection or acute pulmonary embolism;
4. Explicit mechanical complications, including interventricular septum perforation, rupture of papillary muscles and chordae tendineae, or on-going or ruptured left ventricular free walls.
5. Serious cardiogenic shock and do not responding to hypertensive agents;
6. Uncontrolled acute left heart failure or pulmonary edema;
7. Malignant arrhythmias uncontrolled by anti-arrhythmia agents;
8. Bleeding history of cerebral vessels, gastrointestinal tract, respiratory tract, urinary tract or other organs within 1 month;
9. Presence of active hemorrhage at any part of the body (including menstruation);
10. Known hemorrhagic constitution or serious hemostasis and blood coagulation disorders;
11. Current usage of anticoagulants (such as Warfarin or new anticoagulants);
12. . Serious hepatorenal dysfunction [ATL≥5 ULN (upper limit of normal), Cr>134μmol/L (2mg%) or eGFR<45ml/min/1.73m2];
13. Serious chronic obstructive pulmonary disease (COPD) or respiratory failure;
14. . Severe infection:
15. . Very weak or frailty;
16. . Neuropsychiatric system diseases;
17. . Malignancies;
18. . Other pathophysiological conditions with expected survival time <1 year;
19. Allergy to the ingredients of this investigational drug;
20. Women who are in pregnancy or nursery;
21. Participation in clinical study of other traditional Chinese medicine (TCM);
22. Unsuitability to participate in this study due to other diseases.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3796 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
MACCE | 30-day
  30-day incidence of composite endpoint events comprising MACCE (including cardiovascular death, myocardial re-infarction, emergency coronary revascularization and cerebral stroke)

SECONDARY OUTCOMES:
Revascularization | 30-day
  Incidence of revascularization of the primary endpoints
Cerebral stroke | 30-day
  Incidence of cerebral stroke of the primary endpoints
STEMI | 30-day
  30-day incidence of severe complications of STEMI including cardiogenic shock, heart failure, mechanical complications and malignant arrhythmias.
The incidence of bleeding in BARC（Bleeding Academic Research Committee Bleeding Standard） III and V | 30-day
  The incidence of bleeding in BARC（Bleeding Academic Research Committee Bleeding Standard） III and V at 30-day between 0-30%.
MACCE | 1 year
  1-year incidence of composite endpoints comprising MACCE (including cardiovascular death, myocardial re-infarction, emergency coronary revascularization and cerebral stroke), re-hospitalization due to heart failure, in-stent thrombosis and major bleeding (BARC grade III and V), and the incidence of each primary endpoint event.
In-stent restenosis | 1 year
  1-year incidence of In-stent restenosis
All-cause mortality rate at 1 year | 1 year
  Symptoms improved after treatment. Evaluate all-cause mortality rate at 1 year.
Myocardial reperfusion and no-reflow | 2 hours, 24 hours and 7 days
  Evaluation of Myocardial reperfusion and no-reflow: resolution of elevated ST-segment in ECG and incidence of no-reflow at 2h, 24h and 7 days after reperfusion therapy.

OTHER OUTCOMES:
Total white cell count | 7 days, 1 month, 6 months and 1 year after medication
  Normal value: 4-10, unit: 109/L.Check at 7 days, 1 month, 6 months and 1 year to see if it is within the normal range.
Red blood cell | 7 days, 1 month, 6 months and 1 year after medication
  Normal value: 3.5-5, unit: 1012/L.Check at 7 days, 1 month, 6 months and 1 year to see if it is within the normal range.
Hemoglobin | 7 days, 1 month, 6 months and 1 year after medication
  Normal value: 110-150, unit: g/L.Check at 7 days, 1 month, 6 months and 1 year to see if it is within the normal range.
Blood platelet count | 7 days, 1 month, 6 months and 1 year after medication
  Normal value: 100-300, unit: 109/L.Check at 7 days, 1 month, 6 months and 1 year to see if it is within the normal range.

CONTACTS AND LOCATIONS:
Overall Officials: Yue-Jin Yang, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (7):
- China (7):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Beijing Aerospace General Hospital, Beijing, Beijing Municipality
  - Beijing Renhe Hospital, Beijing, Beijing Municipality
  - Harrison International Peace Hospital, Hengshui, Hebei
  - Henan Provincial Peoples Hospital, Zhengzhou, Henan
  - Taian City Central Hospital, Tai’an, Shandong
  - First Teaching Hospital of Tianjin University of TCM, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Li X, Chen G, Xian Y, Zhang H, Wu Y, Yang Y, Wu J, Wang C, He S, Wang Z, Wang Y, Wang Z, Liu H, Wang X, Zhang M, Zhang J, Li J, An T, Guan H, Li L, Shang M, Yao C, Han Y, Zhang B, Gao R, Peterson ED; CTS-AMI Investigators. Traditional Chinese Medicine Compound (Tongxinluo) and Clinical Outcomes of Patients With Acute Myocardial Infarction: The CTS-AMI Randomized Clinical Trial. JAMA. 2023 Oct 24;330(16):1534-1545. doi: 10.1001/jama.2023.19524. PMID 37874574